CLINICAL TRIAL: NCT04942912
Title: Effect of Enzyme Replacement Therapy in Patients With Juvenile-Onset Pompe Disease: a Long-term Observational Study
Brief Title: Effect of Enzyme Replacement Therapy in Patients With Juvenile-onset Pompe Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, FEILLET François, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI280
Record Dates: First submitted 2021-04-17; First posted 2021-06-29 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Pompe's Disease Juvenile Onset
Keywords: no cardiomyopathy at diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- French patients with juvenile Pompe disease: We aim to include all French patients with juvenile Pompe disease (maltase acid deficiency without cardiomyopathy)

SUMMARY:
Pompe disease is known as glycogen storage disease type II, an autosomal recessive disease that results from acid alpha-glucosidase (GAA) deficiency leading to lysosomal glycogen accumulation. Patients with classic infantile form have less than 1% of enzyme activity, which explains severe impairment before one year with rapid death without treatment, while later-onset form shows progressive symptoms later in childhood (juvenile form) or adulthood (adult form).

Enzyme replacement therapy (ERT) consists of periodic intravenous infusion of missing GAA produced by the recombinant method. ERT improves significantly the cardiac function and the children's survival in classic infantile form. This therapy has been approved for all patients with Pompe's disease in the United States and the European Union since 2006, but its efficacy was not clear for patients with later-onset form. Recent studies show motor improvement in adult patients, but there is little published data for the juvenile form disease. A separate analysis of juvenile form is justified as patients are still in a developmental stage and show clinical symptoms early in life, may have more severe disease and a different response to ERT. The recommendation is no treatment in the absence of clinical symptoms, but the consensus does not stratify patients into juvenile- or adult-onset form. ERT is an expensive long-term therapy, and its administration every 2 weeks in the hospital is a great limitation for patients. Therefore, an evaluation of the treatment effect in patients with the juvenile form is necessary.

DETAILED DESCRIPTION:
This study includes patients from several hospitals in france. The parameters allowing the evaluation of the respiratory and muscular function are collected.

ELIGIBILITY:
Inclusion Criteria:

* childhood Pompe disease (the first symptoms appear before 18 years old)
* follow-up in France

Exclusion Criteria:

* infantile Pompe disease
* cardiomyopathy at diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study includes the patients who have Pompe disease documented by deficient alpha-glucosidase activity and/or DNA analysis and follow-up in the French referral centers. These patients must be younger than 18 years at diagnosis and not have the infantile form of Pompe disease. The children who have cardiomyopathy at diagnosis are excluded in order to take only juvenile form.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
6-min walk test | Day 1
  Walking distance during 6 minutes
6-min walk test | Through study completion, an average of 1 year
  Walking distance during 6 minutes
Forced vital capacity | Day 1
  Evaluation of respiratory function test
Forced vital capacity | Through study completion, an average of 1 year
  Evaluation of respiratory function test

SECONDARY OUTCOMES:
Blood creatinine kinase level | Day 1
  Biological marker of Pompe disease
Blood creatinine kinase level | Through study completion, an average of 1 year
  Biological marker of Pompe disease
ASAT | Day 1
  Biological markers of tPompe Disease
ASAT | Through study completion, an average of 1 year
  Biological markers of tPompe Disease
ALAT | Day 1
  Biological markers of tPompe Disease
ALAT | Through study completion, an average of 1 year
  Biological markers of tPompe Disease

CONTACTS AND LOCATIONS:
Overall Officials: François FEILLET, MD, PHD, Principal Investigator — Children's Hospital - CHRU de Nancy, France
Locations (1):
- Children's Hospital - CHRU de Nancy, Nancy, France